CLINICAL TRIAL: NCT01229449
Title: A Double-blind, 5 Parallel-group, Placebo-controlled, Randomised, Single Dose, 3-site Study to Compare the Analgesic Efficacy and Tolerability of a Combination of Ibuprofen 400 mg Plus Paracetamol 1000 mg; a Combination of Ibuprofen 200 mg Plus Paracetamol 500 mg; a Combination of Ibuprofen 400 mg Plus Codeine 25.6 mg (Nurofen Plus®); a Combination of Paracetamol 1000 mg Plus Codeine 30 mg (Panadeine® Extra) in Postoperative Adult Dental Pain Following Third Molar Extraction.
Brief Title: Ibuprofen/Acetaminophen Versus Nurofen Plus® and Panadeine® Extra Dental Pain Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Collaborators: Premier Research (Other); Aptuit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL0811
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-08

CONDITIONS: Post-operative Pain
Keywords: Dental pain; Ibuprofen; Acetaminophen; Nurofen Plus®; Panadeine® Extra; Paracetamol
MeSH Terms: conditions — Pain, Postoperative; Toothache | interventions — Ibuprofen; Acetaminophen; Codeine; acetaminophen, codeine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ibuprofen/acetaminophen (lower dose) (Experimental): One tablet of ibuprofen 200 mg plus acetaminophen 500 mg and one placebo tablet
  Interventions: Drug: Ibuprofen/acetaminophen
- Ibuprofen/acetaminophen (higher dose) (Experimental): Two tablets of ibuprofen 200 mg plus acetaminophen 500 mg
  Interventions: Drug: Ibuprofen/acetaminophen (higher dose)
- Nurofen Plus® (Active Comparator): Two tablets ibuprofen 200mg plus codeine 12.8mg (Nurofen Plus®)
  Interventions: Drug: Nurofen Plus®
- Panadeine® Extra (Active Comparator): Two tablets acetaminophen 500 mg plus codeine 15 mg (Panadeine® Extra)
  Interventions: Drug: Panadeine® Extra
- Placebo (Placebo Comparator): Two placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen/acetaminophen — One tablet of ibuprofen 200 mg plus acetaminophen 500 mg and one placebo tablet, single dose taken orally with 300 ml water
  Other Names: Ibuprofen/paracetamol (lower dose)
  Arms: Ibuprofen/acetaminophen (lower dose)
Drug: Ibuprofen/acetaminophen (higher dose) — Two tablets of ibuprofen 200 mg plus acetaminophen 500 mg, single dose taken orally with 300 ml water
  Other Names: Ibuprofen/Paracetamol
  Arms: Ibuprofen/acetaminophen (higher dose)
Drug: Nurofen Plus® — Two tablets ibuprofen 200mg plus codeine 12.8mg (Nurofen Plus®), single dose taken orally with 300 ml water
  Other Names: Ibuprofen/Codeine
  Arms: Nurofen Plus®
Drug: Panadeine® Extra — Two tablets acetaminophen 500 mg plus codeine 15 mg (Panadeine® Extra), single dose taken orally with 300 ml water
  Other Names: Acetaminophen/codeine; Paracetamol/codeine
  Arms: Panadeine® Extra
Drug: Placebo — Two placebo tablets, single dose taken orally with 300 ml water
  Arms: Placebo

SUMMARY:
The objective is to assess the efficacy and tolerability of a combination of 400 mg ibuprofen plus 1000 mg acetaminophen, 200 mg ibuprofen plus 500 mg acetaminophen compared with Nurofen Plus® and Panadeine® Extra.

DETAILED DESCRIPTION:
RB has developed a fixed-dose combination of ibuprofen and acetaminophen (paracetamol). Since the pharmacological actions of ibuprofen and acetaminophen (paracetamol) differ in their site and mode of action, the combination would be expected to be more effective than either active alone, given that pain is multi-factorial with different mediators.

The purpose of this study was to compare the efficacy and tolerability of ibuprofen/acetaminophen (paracetamol) combination with leading market analgesics.

The efficacy and tolerability was assessed in terms of total analgesic effect, peak analgesic effect, onset and duration of action and the subject's overall assessment of the study medication.

ELIGIBILITY:
Main Inclusion Criteria:

Experiencing moderate to severe pain after extraction of impacted third molars

Main Exclusion Criteria:

Any ongoing painful condition other than that associated with the current third molar surgery that could significantly interfere with the subject's suitability Any condition that would render the subject unsuitable to receive an NSAID, acetaminophen or codeine

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Daniels, Principal Investigator — Premier Research Group Inc
Locations (1):
- Premier Research, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in three centres, Salt Lake City (243 subjects randomised), San Marcos (229 subjects randomised) and Austin (206 subjects randomised)
Pre-assignment Details: A total of 678 subjects were randomised into the study.173 subjects received ibuprofen 200 mg + paracetamol 500 mg, 169 subjects received Nurofen Plus®, 168 subjects received ibuprofen 400 mg + paracetamol 1000 mg, 113 subjects received Panadeine® Extra and 55 subjects received placebo.
Groups:
- Ibuprofen 200mg + Paracetamol 500mg (Lower Dose): One tablet of ibuprofen 200 mg plus acetaminophen 500 mg and one placebo tablet by mouth (single dose)
- Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose): Two tablets of ibuprofen 200 mg plus two tablets of acetaminophen 500 mg by mouth (single dose)
- Nurofen Plus®: Two tablets ibuprofen 200 mg plus codeine 12.8 mg (Nurofen Plus®) by mouth (single dose)
- Panadeine® Extra: Two tablets acetaminophen 500 mg plus codeine 15 mg (Panadeine® Extra) by mouth (single dose)
- Placebo: Two placebo tablets by mouth
Period: Overall Study
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Started | 173 | 168 | 169 | 113 | 55
Completed | 172 | 164 | 167 | 112 | 54
Not Completed | 1 | 4 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ibuprofen 200mg + Paracetamol 500mg (Lower Dose): One tablet of ibuprofen 200 mg plus acetaminophen 500 mg and one placebo tablet by mouth
- Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose): Two tablets of ibuprofen 200 mg plus acetaminophen 500 mg by mouth
- Nurofen Plus®: Two tablets ibuprofen 200mg plus codeine 12.8mg (Nurofen Plus®) by mouth
- Panadeine® Extra: Two tablets acetaminophen 500 mg plus codeine 15 mg (Panadeine® Extra) by mouth
- Total: Total of all reporting groups
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo | Total
Number analyzed (Participants) | 173 | 168 | 169 | 113 | 55 | 678
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.2 (3.3) | 19.8 (3.2) | 20.1 (3.4) | 19.7 (3.3) | 19.8 (3.6) | 20.0 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 100 | 101 | 68 | 33 | 407
  Male | 68 | 68 | 68 | 45 | 22 | 271
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 0 | 0 | 3
  Asian | 3 | 4 | 7 | 1 | 2 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 1 | 0 | 3
  Black or African American | 4 | 4 | 2 | 3 | 2 | 15
  White | 165 | 158 | 154 | 107 | 51 | 635
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 3 | 1 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 173 | 168 | 169 | 113 | 55 | 678
Weight [Mean (Standard Deviation); unit: kg] | 68.1 (14.5) | 69.0 (15.2) | 68.8 (15.3) | 70.8 (16.1) | 71.0 (18.7) | 69.2 (15.5)
Height [Mean (Standard Deviation); unit: cm] | 168.5 (10.0) | 169.3 (10.1) | 169.5 (9.8) | 168.5 (9.7) | 168.7 (9.5) | 168.9 (9.9)
Drink alcohol [Number; unit: participants] | 63 | 61 | 61 | 36 | 15 | 236
Former smoker [Number; unit: participants] | 27 | 23 | 20 | 13 | 9 | 92
Current smoker [Number; unit: participants] | 16 | 16 | 16 | 14 | 5 | 67
Used drugs of abuse [Number; unit: participants] | 32 | 31 | 37 | 18 | 8 | 126

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Area Under the Curve (AUC) of Pain Intensity and Relief Scores (SPRID)
Description: SPRID 0-12h: Sum of pain intensity difference (PID) and the pain relief (PR) score over the twelve-hour follow-up period. Score range: 0mm = No pain and 100mm = Worst pain. This was calculated as the area under the curve (AUC) using the method of linear trapezoids assuming that the baseline assessment took place at time zero.
  Pain intensity (PI) was measured by pain assessment questionnaire, where subject tick the appropriate box in a 4-point ordinal scale ranging from 0 = No pain, 1 = Mild pain, 2 = Moderate pain, and 3 = Severe pain, in response to the question 'What is your pain level at this time?'
  Total Pain Relief (TOTPAR) was measured using pain assessment diary, where subject tick the appropriate box on a 5-point Ordinal Rating Scale: 0 = None, 1 = A Little, 2 = Some, 3 = A Lot, and 4 = Complete, in response to the question 'How much relief have you had from your starting pain?'
Time Frame: 0 (baseline), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: Intention-to-treat (ITT) population includes all randomized subjects who took the study medication, completed the baseline efficacy assessments and had at least one post-baseline assessment. Any subjects with treatment administration errors were analyzed according to the treatment to which they were randomized.
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Number analyzed (Participants) | 173 | 168 | 169 | 113 | 55
units on a scale*hour | 2.68 (1.59) | 3.30 (1.67) | 2.62 (1.73) | 1.93 (1.51) | 0.54 (1.37)
Statistical Analysis 1: Comparison: Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) vs Placebo; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) vs Panadeine® Extra; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) vs Nurofen Plus®; Test type: Superiority; p = 0.0001, ANOVA
Statistical Analysis 4: Comparison: Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) vs Panadeine® Extra; Test type: Superiority; p = 0.0001, ANOVA
Statistical Analysis 5: Comparison: Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) vs Nurofen Plus®; Test type: Superiority; p = 0.72, ANOVA
Statistical Analysis 6: Comparison: Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) vs Placebo; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 7: Comparison: Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) vs Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose); Test type: Superiority; p = 0.0005, ANOVA
Statistical Analysis 8: Comparison: Nurofen Plus® vs Panadeine® Extra; Test type: Superiority; p = 0.0005, ANOVA
Statistical Analysis 9: Comparison: Nurofen Plus® vs Placebo; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 10: Comparison: Panadeine® Extra vs Placebo; Test type: Superiority; p < 0.0001, ANOVA

2. Secondary Outcome: Change From Baseline in AUC (0-8h) of SPRID
Description: SPRID 0-8h: Sum of pain intensity difference (PID) and the pain relief (PR) score over the twelve-hour follow-up period. Score range: 0 mm = No pain and 100 mm = Worst pain. This was calculated as the area under the curve (AUC) using the method of linear trapezoids assuming that the baseline assessment took place at time zero.
  Pain intensity (PI) was measured by pain assessment questionnaire, where subject tick the appropriate box in a 4-point ordinal scale ranging from 0 = No pain, 1 = Mild pain, 2 = Moderate pain, and 3 = Severe pain, in response to the question 'What is your pain level at this time?'
  Total Pain Relief (TOTPAR) was measured using pain assessment diary, where subject tick the appropriate box on a 5-point Ordinal Rating Scale: 0 = None, 1 = A Little, 2 = Some, 3 = A Lot, and 4 = Complete, in response to the question 'How much relief have you had from your starting pain?'
Time Frame: 0 (baseline), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Number analyzed (Participants) | 173 | 168 | 169 | 113 | 55
units on a scale*hour
  0-4h | 3.65 (1.60) | 3.95 (1.52) | 3.44 (1.72) | 3.19 (1.61) | 0.61 (1.26)
  0-6h | 3.66 (1.68) | 4.06 (1.64) | 3.45 (1.82) | 2.86 (1.62) | 0.60 (1.32)
  0-8h | 3.39 (1.71) | 3.91 (1.69) | 3.22 (1.85) | 2.48 (1.57) | 0.57 (1.31)

3. Secondary Outcome: Change From Baseline in AUC for Pain Intensity Difference Scores (SPID)
Description: Sum of Pain Intensity Difference (SPID) was calculated as the area under the curve (AUC) using the method of linear trapezoids assuming that the baseline assessment took place at time zero. Score range: 0mm = No pain and 100mm = Worst pain. Pain intensity (PI) was measured by pain assessment questionnaire, where subject tick the appropriate box in a 4-point ordinal scale ranging from 0 = No pain, 1 = Mild pain, 2 = Moderate pain, and 3 = Severe pain, in response to the question 'What is your pain level at this time?'
Time Frame: 0-4, 0-6, 0-8 and 0-12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Number analyzed (Participants) | 173 | 168 | 169 | 113 | 55
units on a scale*hour
  0-4h | 1.32 (0.73) | 1.46 (0.72) | 1.23 (0.75) | 1.13 (0.70) | 0.18 (0.53)
  0-6h | 1.32 (0.74) | 1.50 (0.75) | 1.23 (0.76) | 1.01 (0.67) | 0.19 (0.53)
  0-8h | 1.21 (0.73) | 1.43 (0.75) | 1.14 (0.75) | 0.87 (0.63) | 0.19 (0.53)
  0-12h | 0.94 (0.64) | 1.18 (0.69) | 0.91 (0.67) | 0.67 (0.57) | 0.19 (0.56)

4. Secondary Outcome: Change From Baseline in AUC of Pain Relief Scores (TOTPAR)
Description: Total pain relief (TOTPAR) was measured using pain assessment diary where subject tick the appropriate box in response to the question 'How much relief have you had from your starting pain?'
  Pain Relief (PR) was rated on a 5-point Ordinal Rating Scale: 0 = None, 1 = A Little, 2 = Some, 3 = A Lot, and 4 = Complete.
Time Frame: 0-4, 0-6, 0-8 and 0-12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Number analyzed (Participants) | 173 | 168 | 169 | 113 | 55
units on a scale*hour
  0-4h | 2.33 (0.96) | 2.48 (0.90) | 2.20 (1.04) | 2.05 (1.00) | 0.42 (0.77)
  0-6h | 2.34 (1.02) | 2.56 (0.98) | 2.22 (1.12) | 1.85 (1.03) | 0.41 (0.82)
  0-8h | 2.18 (1.05) | 2.48 (1.03) | 2.08 (1.15) | 1.61 (1.01) | 0.38 (0.81)
  0-12h | 1.73 (1.01) | 2.12 (1.06) | 1.70 (1.11) | 1.27 (0.98) | 0.34 (0.82)

5. Secondary Outcome: Change From Baseline in AUC of Individual Reading Pain Intensity and Relief Scores (SPRID)
Description: as for outcome 1
Time Frame: 15, 30, 45, 60, 90 minutes and 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Number analyzed (Participants) | 173 | 168 | 169 | 113 | 55
units on a scale
  15 minutes | 1.12 (1.21) | 1.29 (1.38) | 0.78 (1.22) | 1.01 (1.40) | 0.29 (0.74)
  30 minutes | 2.49 (1.63) | 2.79 (1.62) | 2.08 (1.71) | 2.62 (1.83) | 0.58 (1.13)
  45 minutes | 3.20 (1.72) | 3.52 (1.64) | 2.92 (1.84) | 3.39 (1.80) | 0.65 (1.38)
  60 minutes | 3.71 (1.83) | 4.04 (1.66) | 3.49 (1.98) | 3.81 (1.83) | 0.71 (1.49)
  90 minutes | 4.12 (1.82) | 4.44 (1.69) | 3.92 (2.06) | 3.96 (1.77) | 0.60 (1.56)
  2 hours | 4.28 (1.95) | 4.51 (1.80) | 4.17 (2.14) | 3.91 (1.90) | 0.67 (1.43)
  3 hours | 4.18 (2.06) | 4.53 (1.95) | 4.02 (2.14) | 3.31 (2.13) | 1.66 (0.00)
  4 hours | 4.08 (2.09) | 4.46 (2.09) | 3.78 (2.31) | 2.79 (2.21) | 0.64 (1.65)
  5 hours | 3.77 (2.21) | 4.36 (2.12) | 3.52 (2.40) | 2.23 (2.20) | 0.60 (1.59)
  6 hours | 3.06 (2.34) | 3.98 (2.24) | 2.98 (2.47) | 1.70 (2.16) | 0.53 (1.56)
  7 hours | 2.56 (2.37) | 3.51 (2.40) | 2.54 (2.50) | 1.31 (2.00) | 0.45 (1.45)
  8 hours | 2.09 (2.31) | 2.79 (2.49) | 2.08 (2.38) | 1.02 (1.92) | 0.40 (1.30)
  9 hours | 1.57 (2.20) | 2.53 (2.47) | 1.68 (2.20) | 0.91 (1.87) | 0.47 (1.59)
  10 hours | 1.21 (2.02) | 2.04 (2.34) | 1.30 (2.06) | 0.81 (1.84) | 0.49 (1.62)
  11 hours | 0.90 (1.83) | 1.63 (2.24) | 1.12 (2.02) | 0.76 (1.77) | 0.49 (1.62)
  12 hours | 0.69 (1.64) | 1.34 (2.14) | 0.96 (1.85) | 0.74 (1.76) | 0.49 (1.62)

6. Secondary Outcome: Individual Pain Intensity Differences (Ordinal)
Description: Pain intensity (PI) was measured by pain assessment questionnaire where subject tick the appropriate box in response to the question 'What is your pain level at this time?'
  PI measured using a 4-point ordinal scale: 0 = No pain, 1 = Mild pain, 2 = Moderate pain, and 3 = Severe pain.
Time Frame: 15, 30, 45, 60, 90 minutes and 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Number analyzed (Participants) | 173 | 168 | 169 | 113 | 55
units on a scale
  15 minutes | 0.40 (0.57) | 0.46 (0.64) | 0.23 (0.58) | 0.31 (0.64) | 0.09 (0.40)
  30 minutes | 0.94 (0.76) | 1.03 (0.74) | 0.73 (0.80) | 0.95 (0.83) | 0.15 (0.56)
  45 minutes | 1.14 (0.76) | 1.27 (0.76) | 1.04 (0.80) | 1.19 (0.83) | 0.16 (0.63)
  60 minutes | 1.31 (0.85) | 1.48 (0.79) | 1.24 (0.87) | 1.35 (0.85) | 0.22 (0.79)
  90 minutes | 1.49 (0.83) | 1.61 (0.84) | 1.40 (0.92) | 1.42 (0.83) | 0.11 (0.81)
  2 hours | 1.54 (0.89) | 1.69 (0.87) | 1.52 (0.94) | 1.41 (0.84) | 0.24 (0.54)
  3 hours | 1.54 (0.91) | 1.70 (0.89) | 1.46 (0.93) | 1.19 (0.87) | 0.22 (0.66)
  4 hours | 1.49 (0.91) | 1.68 (0.94) | 1.36 (0.95) | 0.96 (0.90) | 0.24 (0.64)
  5 hours | 1.35 (0.93) | 1.60 (0.93) | 1.24 (0.96) | 0.79 (0.88) | 0.22 (0.63)
  6 hours | 1.07 (0.93) | 1.44 (0.93) | 1.04 (0.95) | 0.58 (0.82) | 0.20 (0.62)
  7 hours | 0.89 (0.93) | 1.22 (0.98) | 0.88 (0.96) | 0.44 (0.74) | 0.18 (0.61)
  8 hours | 0.71 (0.89) | 0.96 (0.96) | 0.72 (0.89) | 0.33 (0.71) | 0.16 (0.54)
  9 hours | 0.53 (0.80) | 0.86 (0.94) | 0.55 (0.80) | 0.29 (0.68) | 0.20 (0.68)
  10 hours | 0.40 (0.74) | 0.67 (0.87) | 0.43 (0.75) | 0.27 (0.67) | 0.20 (0.68)
  11 hours | 0.27 (0.64) | 0.52 (0.80) | 0.36 (0.73) | 0.24 (0.63) | 0.20 (0.68)
  12 hours | 0.21 (0.57) | 0.42 (0.78) | 0.30 (0.63) | 0.25 (0.63) | 0.20 (0.68)

7. Secondary Outcome: Individual Pain Intensity Differences Visual Analogue Scale (VAS)
Description: Pain Intensity (PI) VAS was measured using a horizontal 100-mm VAS ranging 0 mm = 'No Pain' as the left anchor and 100 mm = 'Worst Pain' as the right anchor, labelled by the subject marking the VAS line in the pain assessment questionnaire in response to the instruction 'Please indicate with a line on the scale below your pain at this time.'
Time Frame: 15, 30, 45, 60, 90 minutes and 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Number analyzed (Participants) | 173 | 168 | 169 | 113 | 55
units on a scale
  15 minutes | 9.0 (13.7) | 10.5 (16.3) | 4.5 (14.1) | 8.7 (16.6) | 0.4 (13.1)
  30 minutes | 22.8 (21.4) | 26.2 (21.5) | 17.7 (22.5) | 23.9 (23.9) | 2.2 (16.7)
  45 minutes | 32.5 (23.8) | 37.5 (24.0) | 28.3 (25.7) | 34.3 (25.7) | 0.9 (18.8)
  60 minutes | 40.3 (25.5) | 46.3 (24.4) | 36.6 (28.7) | 41.5 (27.1) | 1.8 (19.3)
  90 minutes | 48.3 (25.8) | 52.5 (24.8) | 43.7 (28.2) | 44.6 (25.9) | 0.9 (22.6)
  2 hours | 50.6 (26.6) | 54.9 (25.7) | 47.3 (29.3) | 45.2 (27.9) | 5.0 (18.2)
  3 hours | 51.0 (27.1) | 55.9 (25.5) | 48.0 (29.3) | 38.9 (29.9) | 6.1 (21.3)
  4 hours | 50.2 (27.8) | 55.5 (26.4) | 45.6 (29.9) | 32.9 (29.4) | 7.2 (20.3)
  5 hours | 45.4 (28.7) | 52.8 (26.7) | 42.5 (30.4) | 25.9 (29.2) | 7.2 (19.8)
  6 hours | 36.6 (30.2) | 47.9 (27.8) | 35.6 (30.6) | 18.4 (27.2) | 6.5 (19.7)
  7 hours | 30.9 (30.6) | 41.0 (29.8) | 29.7 (30.8) | 15.4 (25.2) | 5.8 (18.8)
  8 hours | 25.0 (28.9) | 33.8 (30.8) | 24.4 (29.8) | 11.7 (24.4) | 5.1 (17.2)
  9 hours | 17.7 (26.4) | 29.6 (30.3) | 18.4 (27.2) | 10.8 (22.9) | 5.6 (19.4)
  10 hours | 14.1 (25.2) | 23.7 (29.1) | 14.9 (25.3) | 9.7 (22.9) | 6.2 (20.3)
  11 hours | 9.4 (21.2) | 18.7 (27.2) | 12.8 (24.7) | 9.8 (23.2) | 6.2 (20.1)
  12 hours | 8.0 (20.4) | 15.1 (25.5) | 11.0 (22.9) | 9.3 (22.1) | 6.4 (20.8)

8. Secondary Outcome: Change From Baseline in Peak Pain Intensity Difference (Peak PID - Ordinal)
Description: as for outcome 6
Time Frame: 0 (baseline), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Number analyzed (Participants) | 173 | 168 | 169 | 113 | 55
units on a scale | 1.78 (0.83) | 1.93 (0.81) | 1.74 (0.87) | 1.63 (0.77) | 0.60 (0.87)

9. Secondary Outcome: Change From Baseline in Peak Pain Relief (PR)
Description: as for outcome 4
Time Frame: 0 (baseline), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Number analyzed (Participants) | 173 | 168 | 169 | 113 | 55
units on a scale | 3.06 (1.00) | 3.25 (0.89) | 2.98 (1.11) | 2.88 (1.00) | 0.96 (1.15)

10. Secondary Outcome: Subjects' Overall Assessment of the Study Medication Assessed at 12 Hours or Just Before Administration of Rescue Medication
Description: Subject's Overall Assessment measured by subject ticking the appropriate box in response to the question 'How effective do you think the study medication is as a treatment for pain?'
  Subject's Overall Assessment rated on a five-point ordinal scale: 1 = Poor, 2 = Fair, 3 = Good, 4 = Very good, and 5 = Excellent.
Time Frame: At 12 hours
Population: Three subjects from ITT population were excluded from this analysis due to early/late diary assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
Number analyzed (Participants) | 169 | 165 | 167 | 113 | 55
Participants
  1 Poor | 15 | 9 | 15 | 12 | 43
  2 Fair | 16 | 12 | 22 | 19 | 6
  3 Good | 43 | 32 | 40 | 41 | 2
  4 Very good | 72 | 69 | 64 | 34 | 3
  5 Excellent | 23 | 39 | 26 | 7 | 1

ADVERSE EVENTS:
Time Frame: Up to Day 10 (follow-up)
Description: A treatment emergent adverse event is any event commencing within 12 hours of study medication dose.
Arm/Group | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) | Nurofen Plus® | Panadeine® Extra | Placebo
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/168 | 0/169 | 0/113 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/168 | 0/169 | 0/113 | 0/55
Other Adverse Events (participants affected / at risk) | 88/173 | 87/168 | 97/169 | 72/113 | 35/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen 200mg + Paracetamol 500mg (Lower Dose) (N=173) | Ibuprofen 400mg + Paracetamol 1000mg (Higher Dose) (N=168) | Nurofen Plus® (N=169) | Panadeine® Extra (N=113) | Placebo (N=55)
Nausea (Gastrointestinal disorders) | 43 (49) | 33 (36) | 50 (57) | 37 (49) | 18 (19)
Vomiting (Gastrointestinal disorders) | 29 (32) | 30 (34) | 35 (41) | 25 (29) | 13 (13)
Dizziness (Nervous system disorders) | 12 (13) | 15 (16) | 23 (24) | 14 (14) | 3 (4)
Headache (Nervous system disorders) | 19 (23) | 19 (21) | 32 (35) | 21 (30) | 10 (11)
Alveolar osteitis (Infections and infestations) | 8 (8) | 4 (4) | 9 (9) | 3 (3) | 1 (1)
Body temperature increased (Investigations) | 2 (2) | 3 (3) | 9 (9) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator must submit any proposed manuscript to RB for approval prior to submission for publication. No timelines are stated. However, note that the results of this study have already been published.